CLINICAL TRIAL: NCT05593835
Title: Protocol for a Cluster Randomised Trial of a Goal-Oriented Care Approach for Multimorbidity Patients Supported by a Digital Platform
Brief Title: Multimorbidity Management Supported by a Digital Platform
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Administração Regional de Saúde de Lisboa e Vale do Tejo, Portugal (Unknown); Universidade Lusófona de Humanidades e Tecnologias (Other); NOVA Medical School (Other); NOVA School of Science and Technology ı FCT NOVA (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: METHIS_CRTMB2022
Record Dates: First submitted 2022-10-03; First posted 2022-10-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Disease
Keywords: Primary Health Care; Information Management; Research Design; Telemedicine; Digital Health; Patient-Centered Care; Goal-Oriented Care
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Cluster Randomised Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- METHIS Intervention (Experimental): The METHIS intervention will consist of two components. The first component is a Goal-Oriented Care (GOC) Training Program for health professionals. The training program will include the concept of personalised care, methods of goal elation, implications of GOC in healthcare practice, and how METHIS platform can be used to support the application of GOC. The training will be implemented through a blended-learning, continuous education program that will be credited by Nova University of Lisbon. The second component is a GOC information system. This will be the digital platform METHIS, which will be designed to nudge clinicians to adopt a GOC and to encourage patients and caregivers to take an active role in healthcare. The investigators will adapt an existing platform that was developed for a pilot study during the COVID-19 pandemic, that promotes care coordination, optimises disease prioritisation, and patient self-management.
  Interventions: Device: METHIS Platform; Other: Goal-Oriented Care Training Program
- Control (No Intervention): The control group in this trial will be the best usual care, using the standard Electronic Health Records available to the practice. Our understanding of what "best usual care" is for people with multimorbidity is informed by qualitative research in an earlier stage of this project. Our results suggest that healthcare professionals often provide disease-driven care. When faced with multiple healthcare problems, they prioritise based on 1) patient complaints; 2) which condition is less well controlled; or 3) which condition is more likely to adversely impact on patient Health Related-Quality of life. General practitioners and primary care nurses are often not familiar with the Goal-Oriented Care model. However, they already try to implement some of its principles such as identifying patient goals and supporting shared decision making.

INTERVENTIONS:
Device: METHIS Platform — The METHIS platform is a digital healthcare platform, supported by three databases using PostreSQL (based in relational SQL). One of the databases allows adequate internal testing before production. Another database of production (secured with unique access codes) will be created to retrieve data from the practices' and the last database for the research data, where pseudonymised production data can be analysed for research purposes. The platform is integrated (via FCCN Scientific Computation Unit of the Portuguese Fundação para a Ciência e a Tecnologia) with the Software Zoom® to allow encrypted teleconsultations, with a guarantee that each patient connection is unique. The digital platform is web-based, and it can be used in multiple devices.
  Other Names: Goal-Oriented Care Information System; GOC Information System
  Arms: METHIS Intervention
Other: Goal-Oriented Care Training Program — The training program will have three stages: initial face-to-face training, which will happen before the data collection, followed by remote, asynchronous training during a 12-month period, and a final seminar to discuss the results and inquire about the usability of the GOC model and the METHIS platform. The course will be offered to the intervention group one month before the start of patient recruitment, and for the control group at least one month after the end of data collection.
  Other Names: GOC Training Program
  Arms: METHIS Intervention

SUMMARY:
This study aims to assess whether the use of the METHIS digital platform using a patient-centered approach contributes to an improvement in the quality of life, mental health and physical activity of patients with multimorbidity followed up in Primary Health Care. Practices will be randomly allocated between: providing access to consultations through the METHIS platform (intervention) or following patients by the traditional method (control). They will complete questionnaires on quality of life, mental health and report the number of steps taken, at the beginning and end of the study.

DETAILED DESCRIPTION:
A superiority, cluster randomised trial will be conducted at Primary Health Care Practices (1:1 allocation ratio). All public practices in the Lisbon and Tagus Valley Region, Portugal, not involved in a previous pilot trial, will be eligible. The intervention combines a training programme and a customised Information System (METHIS). Both are designed to help clinicians to adopt a Goal-Oriented Care Model approach and to encourage patients and carers to play a more active role in autonomous healthcare.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling people
* aged 50 or older
* with complex multimorbidity (co-occurrence of three or more chronic conditions affecting three or more different body systems)
* with access to an Internet connection and a communication technology device

Exclusion Criteria:

* inability to: provide informed consent, to read or write, inability to access an email or electronic device, even when helped by an informal caregiver

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Participants will be asked to fill in the SF-12 questionnaire at baseline and at 12 months.
  Participants will be asked to fill in the SF-12 questionnaire which generates a physical component score (PCS) and a mental component score (MCS). The primary outcome will be the mean difference in the variation (delta) of the PCS of SF-12 between baseline and 12 months. The SF-12 can be filled in 2-4 minutes, and it is validated for the Portuguese population. Minimum important differences validated across large populations and multiple disease categories are a change in between 2 and 3 points from the population mean of 50.

SECONDARY OUTCOMES:
Mental health status | Participants will complete the HADS-A and HADS-D questionnaire at baseline and at 12 months.
  Participants will be asked to complete the Hospital Anxiety and Depression Scale questionnaire (HADS-A and HADS-D, respectively). The investigators will calculate the mean difference in the variation (delta) in HADS-A and HADS-D between baseline and 12 months. Although HADS was designed for inpatients it was posteriorly validated in the primary care outpatient setting. A minimum important difference of 1.5 has been reported in other chronic disorders.
Physical activity | Participants will wear the SmartBand for 12 months.
  Physical activity will be monitored through the number of steps walked daily. To assess the number of steps per day, a smart band with a triaxial Accelerometer will be used in both arms of the trial. Although traditional step counters use pedometers to detect daily step counts, accelerometers are more accurate and sensitive to lower force accelerations (e.g., slow walking) being considered the current standard for collecting physical activity data. Sedentary older adults and individuals living with disability and chronic illness benefit from a physically active lifestyle, with approximately 4,600- 5,500 daily steps. The lowest median values for steps/day found is in disabled older adults (1214 steps/day) and by people living with COPD (2237 steps/day).
Number of serious adverse events (clinician-reported) | Family physicians will be asked, at 6 and 12 months after randomization, to check the life status of enrolled patients and whether patients in the trial were admitted to a hospital or had a visit to an emergency service since the randomization date.
  These will be the safety outcomes chosen for this trial. In both trial arms, data about patient mortality will be collected and combined with data on occurrence of emergency department visits and hospital admissions as a proxy for serious adverse events. This information is available through the Portuguese common EHR. Due to legal requirements, after death, the information about hospital admissions and other contacts with healthcare organisations ceases to be available to the attending physician.
Number of potentially missed diagnoses (clinician-reported) | Potentially missed diagnoses will be reported 6 months after the intervention phase. In this way a compromise between avoiding recall bias and allowing enough time for a missed diagnosis to become clinically apparent is achieved.
  These will be a second safety outcome. The investigators will ask clinicians in the intervention arm if they are aware of any serious diagnosis that might have been missed due to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Luís V. Lapão, PhD, Principal Investigator — Universidade Nova de Lisboa

IPD SHARING:
Plan to Share IPD: Yes
The complete research dataset will be stored in an encrypted and secure location with the purpose of being accessed for secondary analyses or comparative studies or per request of the patients involved or the Research and Ethics Committee. For legal reasons, the investigators will not disclose the database or grant access for data reproduction. However, processed data may be made available upon request to the research team, with appropriate justification.
Supporting Information: Study Protocol, CSR
Time Frame: After the study ends and for 5 years.
Access Criteria: The trial protocol, the main paper with the trial results and a short paper with the results of the final physician survey will be published in peer-review journals.

REFERENCES:
- [Background] Onder G, Palmer K, Navickas R, Jureviciene E, Mammarella F, Strandzheva M, Mannucci P, Pecorelli S, Marengoni A; Joint Action on Chronic Diseases and Promoting Healthy Ageing across the Life Cycle (JA-CHRODIS). Time to face the challenge of multimorbidity. A European perspective from the joint action on chronic diseases and promoting healthy ageing across the life cycle (JA-CHRODIS). Eur J Intern Med. 2015 Apr;26(3):157-9. doi: 10.1016/j.ejim.2015.02.020. Epub 2015 Mar 18. PMID 25797840
- [Background] Mercer S, Furler J, Moffat K, Fischbacher-Smith D, Sanci LA, World Health Organization, et al. Multimorbidity: Technical Series on Safer Primary Care. Geneva, Switzerland: World Health Organization; 2016
- [Background] Quinaz Romana G, Kislaya I, Salvador MR, Cunha Goncalves S, Nunes B, Dias C. [Multimorbidity in Portugal: Results from The First National Health Examination Survey]. Acta Med Port. 2019 Feb 1;32(1):30-37. doi: 10.20344/amp.11227. Epub 2019 Feb 1. Portuguese. PMID 30753801
- [Background] Amer Nordin A, Mohd Hairi F, Choo WY, Hairi NN. Care Recipient Multimorbidity and Health Impacts on Informal Caregivers: A Systematic Review. Gerontologist. 2019 Sep 17;59(5):e611-e628. doi: 10.1093/geront/gny072. PMID 29982539
- [Background] van der Aa MJ, van den Broeke JR, Stronks K, Plochg T. Patients with multimorbidity and their experiences with the healthcare process: a scoping review. J Comorb. 2017 Jan 27;7(1):11-21. doi: 10.15256/joc.2017.7.97. eCollection 2017. PMID 29090185
- [Background] Fortin M, Lapointe L, Hudon C, Vanasse A, Ntetu AL, Maltais D. Multimorbidity and quality of life in primary care: a systematic review. Health Qual Life Outcomes. 2004 Sep 20;2:51. doi: 10.1186/1477-7525-2-51. PMID 15380021
- [Background] Makovski TT, Schmitz S, Zeegers MP, Stranges S, van den Akker M. Multimorbidity and quality of life: Systematic literature review and meta-analysis. Ageing Res Rev. 2019 Aug;53:100903. doi: 10.1016/j.arr.2019.04.005. Epub 2019 Apr 30. PMID 31048032
- [Background] Marengoni A, von Strauss E, Rizzuto D, Winblad B, Fratiglioni L. The impact of chronic multimorbidity and disability on functional decline and survival in elderly persons. A community-based, longitudinal study. J Intern Med. 2009 Feb;265(2):288-95. doi: 10.1111/j.1365-2796.2008.02017.x. PMID 19192038
- [Background] Boyd CM, Darer J, Boult C, Fried LP, Boult L, Wu AW. Clinical practice guidelines and quality of care for older patients with multiple comorbid diseases: implications for pay for performance. JAMA. 2005 Aug 10;294(6):716-24. doi: 10.1001/jama.294.6.716. PMID 16091574
- [Background] Cairo Notari S, Sader J, Caire Fon N, Sommer JM, Pereira Miozzari AC, Janjic D, Nendaz M, Audetat MC. Understanding GPs' clinical reasoning processes involved in managing patients suffering from multimorbidity: A systematic review of qualitative and quantitative research. Int J Clin Pract. 2021 Sep;75(9):e14187. doi: 10.1111/ijcp.14187. Epub 2021 May 5. PMID 33783098
- [Background] Damarell RA, Morgan DD, Tieman JJ. General practitioner strategies for managing patients with multimorbidity: a systematic review and thematic synthesis of qualitative research. BMC Fam Pract. 2020 Jul 1;21(1):131. doi: 10.1186/s12875-020-01197-8. PMID 32611391
- [Background] Spencer-Bonilla G, Quinones AR, Montori VM; International Minimally Disruptive Medicine Workgroup. Assessing the Burden of Treatment. J Gen Intern Med. 2017 Oct;32(10):1141-1145. doi: 10.1007/s11606-017-4117-8. Epub 2017 Jul 11. PMID 28699060
- [Background] Whitehead L, Palamara P, Allen J, Boak J, Quinn R, George C. Nurses' perceptions and beliefs related to the care of adults living with multimorbidity: A systematic qualitative review. J Clin Nurs. 2022 Oct;31(19-20):2716-2736. doi: 10.1111/jocn.16146. Epub 2021 Dec 6. PMID 34873763
- [Background] Muth C, Blom JW, Smith SM, Johnell K, Gonzalez-Gonzalez AI, Nguyen TS, Brueckle MS, Cesari M, Tinetti ME, Valderas JM. Evidence supporting the best clinical management of patients with multimorbidity and polypharmacy: a systematic guideline review and expert consensus. J Intern Med. 2019 Mar;285(3):272-288. doi: 10.1111/joim.12842. Epub 2018 Dec 10. PMID 30357955
- [Background] Kernick D, Chew-Graham CA, O'Flynn N. Clinical assessment and management of multimorbidity: NICE guideline. Br J Gen Pract. 2017 May;67(658):235-236. doi: 10.3399/bjgp17X690857. No abstract available. PMID 28450343
- [Background] De Maeseneer J, Boeckxstaens P. James Mackenzie Lecture 2011: multimorbidity, goal-oriented care, and equity. Br J Gen Pract. 2012 Jul;62(600):e522-4. doi: 10.3399/bjgp12X652553. No abstract available. PMID 22782000
- [Background] Gonzalez AI GONZALEZ, Schmucker C, Nothacker J, Motschall E, Nguyen TS, Brueckle MS, Blom J, van den Akker M, Rottger K, Wegwarth O, Hoffmann T, Straus SE, Gerlach FM, Meerpohl JJ, Muth C. Health-related preferences of older patients with multimorbidity: an evidence map. BMJ Open. 2019 Dec 15;9(12):e034485. doi: 10.1136/bmjopen-2019-034485. PMID 31843855
- [Background] Mold JW, Blake GH, Becker LA. Goal-oriented medical care. Fam Med. 1991 Jan;23(1):46-51. PMID 2001782
- [Background] Steele Gray C, Grudniewicz A, Armas A, Mold J, Im J, Boeckxstaens P. Goal-Oriented Care: A Catalyst for Person-Centred System Integration. Int J Integr Care. 2020 Nov 4;20(4):8. doi: 10.5334/ijic.5520. PMID 33199976
- [Background] Goncalves-Bradley DC, J Maria AR, Ricci-Cabello I, Villanueva G, Fonhus MS, Glenton C, Lewin S, Henschke N, Buckley BS, Mehl GL, Tamrat T, Shepperd S. Mobile technologies to support healthcare provider to healthcare provider communication and management of care. Cochrane Database Syst Rev. 2020 Aug 18;8(8):CD012927. doi: 10.1002/14651858.CD012927.pub2. PMID 32813281
- [Background] Gagnon MP, Godin G, Gagne C, Fortin JP, Lamothe L, Reinharz D, Cloutier A. An adaptation of the theory of interpersonal behaviour to the study of telemedicine adoption by physicians. Int J Med Inform. 2003 Sep;71(2-3):103-15. doi: 10.1016/s1386-5056(03)00094-7. PMID 14519403
- [Background] Shojania KG, Jennings A, Mayhew A, Ramsay CR, Eccles MP, Grimshaw J. The effects of on-screen, point of care computer reminders on processes and outcomes of care. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD001096. doi: 10.1002/14651858.CD001096.pub2. PMID 19588323
- [Background] Lamprell K, Tran Y, Arnolda G, Braithwaite J. Nudging clinicians: A systematic scoping review of the literature. J Eval Clin Pract. 2021 Feb;27(1):175-192. doi: 10.1111/jep.13401. Epub 2020 Apr 27. PMID 32342613
- [Background] Kraef C, van der Meirschen M, Free C. Digital telemedicine interventions for patients with multimorbidity: a systematic review and meta-analysis. BMJ Open. 2020 Oct 13;10(10):e036904. doi: 10.1136/bmjopen-2020-036904. PMID 33051232
- [Background] Pascual-de la Pisa B, Palou-Lobato M, Marquez Calzada C, Garcia-Lozano MJ. [Effectiveness of interventions based on telemedicine on health outcomes in patients with multimorbidity in Primary Care: A systematic review]. Aten Primaria. 2020 Dec;52(10):759-769. doi: 10.1016/j.aprim.2019.08.004. Epub 2019 Dec 5. Spanish. PMID 31813545
- [Background] Berntsen G, Strisland F, Malm-Nicolaisen K, Smaradottir B, Fensli R, Rohne M. The Evidence Base for an Ideal Care Pathway for Frail Multimorbid Elderly: Combined Scoping and Systematic Intervention Review. J Med Internet Res. 2019 Apr 22;21(4):e12517. doi: 10.2196/12517. PMID 31008706
- [Background] Lapao LV, Peyroteo M, Maia M, Seixas J, Gregorio J, Mira da Silva M, Heleno B, Correia JC. Implementation of Digital Monitoring Services During the COVID-19 Pandemic for Patients With Chronic Diseases: Design Science Approach. J Med Internet Res. 2021 Aug 26;23(8):e24181. doi: 10.2196/24181. PMID 34313591
- [Background] Kastner M, Hayden L, Wong G, Lai Y, Makarski J, Treister V, Chan J, Lee JH, Ivers NM, Holroyd-Leduc J, Straus SE. Underlying mechanisms of complex interventions addressing the care of older adults with multimorbidity: a realist review. BMJ Open. 2019 Apr 3;9(4):e025009. doi: 10.1136/bmjopen-2018-025009. PMID 30948577
- [Background] Quinaz Romana G, Kislaya I, Cunha Goncalves S, Salvador MR, Nunes B, Matias Dias C. Healthcare use in patients with multimorbidity. Eur J Public Health. 2020 Feb 1;30(1):16-22. doi: 10.1093/eurpub/ckz118. PMID 31978229
- [Background] Broeiro, P. (2015). Multimorbilidade e comorbilidade: duas perspectivas da mesma realidade. Revista Portuguesa De Medicina Geral E Familiar, 31(3), 150-60.
- [Background] Peyroteo M. O sistema de informação e o modelo de orientação na prestação de cuidados de saúde em pacientes com multimorbilidade numa unidade de saúde familiar em Lisboa: uma perspetiva dos profissionais de saúde Instituto de Higiene Tropical, Universidade NOVA de Lisboa; 2020. Available from: https://run.unl.pt/handle/10362/116922
- [Background] Smith SM, Wallace E, Salisbury C, Sasseville M, Bayliss E, Fortin M. A Core Outcome Set for Multimorbidity Research (COSmm). Ann Fam Med. 2018 Mar;16(2):132-138. doi: 10.1370/afm.2178. PMID 29531104
- [Background] Cheung AS, de Rooy C, Hoermann R, Lim Joon D, Zajac JD, Grossmann M. Quality of life decrements in men with prostate cancer undergoing androgen deprivation therapy. Clin Endocrinol (Oxf). 2017 Mar;86(3):388-394. doi: 10.1111/cen.13249. Epub 2016 Nov 2. PMID 27696495
- [Background] Gonzalez-Ortega M, Gene-Badia J, Kostov B, Garcia-Valdecasas V, Perez-Martin C. Randomized trial to reduce emergency visits or hospital admissions using telephone coaching to complex patients. Fam Pract. 2017 Apr 1;34(2):219-226. doi: 10.1093/fampra/cmw119. PMID 27920119
- [Background] Bunevicius A, Peceliuniene J, Mickuviene N, Valius L, Bunevicius R. Screening for depression and anxiety disorders in primary care patients. Depress Anxiety. 2007;24(7):455-60. doi: 10.1002/da.20274. PMID 17117433
- [Background] Puhan MA, Frey M, Buchi S, Schunemann HJ. The minimal important difference of the hospital anxiety and depression scale in patients with chronic obstructive pulmonary disease. Health Qual Life Outcomes. 2008 Jul 2;6:46. doi: 10.1186/1477-7525-6-46. PMID 18597689
- [Background] Corder K, Brage S, Ekelund U. Accelerometers and pedometers: methodology and clinical application. Curr Opin Clin Nutr Metab Care. 2007 Sep;10(5):597-603. doi: 10.1097/MCO.0b013e328285d883. PMID 17693743
- [Background] Tudor-Locke C, Craig CL, Aoyagi Y, Bell RC, Croteau KA, De Bourdeaudhuij I, Ewald B, Gardner AW, Hatano Y, Lutes LD, Matsudo SM, Ramirez-Marrero FA, Rogers LQ, Rowe DA, Schmidt MD, Tully MA, Blair SN. How many steps/day are enough? For older adults and special populations. Int J Behav Nutr Phys Act. 2011 Jul 28;8:80. doi: 10.1186/1479-5868-8-80. PMID 21798044
- [Background] Arvidsson D, Fridolfsson J, Borjesson M. Measurement of physical activity in clinical practice using accelerometers. J Intern Med. 2019 Aug;286(2):137-153. doi: 10.1111/joim.12908. Epub 2019 Apr 16. PMID 30993807
- [Background] Richardson, S. and D. Mackinnon. (2017). Left to their own Devices? Privacy Implications of Wearable Technology in Canadian Workplaces. Surveillance Studies Centre. Available at: https://www.surveillance-studies.ca/sites/sscqueens.org/files/left_to_their_own_devices.pdf
- [Background] Evenson KR, Goto MM, Furberg RD. Systematic review of the validity and reliability of consumer-wearable activity trackers. Int J Behav Nutr Phys Act. 2015 Dec 18;12:159. doi: 10.1186/s12966-015-0314-1. PMID 26684758
- [Result] Johnson EJ, Goldstein D. Medicine. Do defaults save lives? Science. 2003 Nov 21;302(5649):1338-9. doi: 10.1126/science.1091721. No abstract available. PMID 14631022
- [Derived] Gil Conde M, Peyroteo M, Maria A, Maia MR, Gregorio J, Paulo MS, Alves M, Papoila AL, Lapao LV, Heleno B. Protocol for a cluster randomised trial of a goal-oriented care approach for multimorbidity patients supported by a digital platform. BMJ Open. 2023 Nov 17;13(11):e070044. doi: 10.1136/bmjopen-2022-070044. PMID 37977860